CLINICAL TRIAL: NCT00694824
Title: Traditional and Not Traditional Risk Factors in Appearance and Progression of Vascular Calcification in Haemodialysis Patients.
Brief Title: Vascular Calcification's Risk Factors in Haemodialysis Patients
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: University of Bologna (Other)
Responsible Party: Professor Sergio Stefoni, Nephrology Dialysis and Renal Transplantation Unit
Other Study IDs: CVAS-INT-02
Record Dates: First submitted 2008-06-09; First posted 2008-06-11 (Estimated); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Chronic Kidney Failure; Inflammation; Vascular Calcification
Keywords: Coronary artery calcification; calcium score; (TGF) b1,; fetuin A; osteoprotegerin (OPG); fibroblast growth factor (FGF) 23,; matrix gla protein (MGP); hemodialysis patients
MeSH Terms: conditions — Kidney Failure, Chronic; Inflammation; Vascular Calcification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — For each patient a blood sample was drawn to check the basal values of hemoglobin, hematocrit, folates, vitamin B12, C reactive protein, PTH, calcium, phosphorus, albumin, alkaline phosphatase, total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides, uric acid, fibrinogen, homocysteine. To better understand the mineral methabolism TGFb1, fetuin A, OPG, FGF 23, OPN and MGP will be checked. The values for each patient will be the median of 4 determinations, each sample was drawn before the midweek dialysis session.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A

SUMMARY:
A not randomized , cross sectional study will be done to determine the possible association of coronary artery calcification (CAC) score assessed by multirow spiral computed tomography (MSCT) with specific and non specific uremic factor of vascular calcification.

DETAILED DESCRIPTION:
Cardiovascular diseases (CVD) are the main causes of death and hospitalization in patients affected by ESRD . The risk of death from CVD is already detectable in the early steps of chronic renal failure and it is from 20 to 30 times higher than in the general population. In ESRD patients the traditional risk factors for CVD do not offer a satisfactory explanation for such high mortality and morbidity rate. Among them, calcium-phosphate imbalance, inflammation, dialysis age, anaemia, hyperhomocysteinemia, oxidative stress, malnutrition, high lipoprotein levels and endothelial dysfunction have been considered (4).

Recently more attention has been paid to calcium phosphate imbalance involved either in the presence or the progression of vascular calcification (VC) in ESRD patients. Multiple factors have been noticed to contribute to VC other than mineral metabolism: the use of calcium-based phosphate binders, diabetes, aging, inflammation, cytokines and BMI.

Indeed it is now believed that arterial calcification is an active process that involves the phenotypic transformation of vascular smooth muscle cells (VSMC) into bone-forming osteoblast (ob)-like cells that are capable of expressing and/or release bone matrix proteins that are necessary to support the calcification process: OPG, RANKL, OPN, fetuin A and MGP. Several stimuli, first of all mineral changes have been shown to induce o modulate this phenotypic transformation. Indeed the expression and secretion of the above-mentioned proteins is regulated by several molecules such as TGF β, peroxisome proliferator-activated receptors (PPAR) γ, tumor necrosis factor (TNF) α.

Calcification develops at two sites in arterial wall, the intima and the media layers: 1)intimal calcification is frequent in advanced stages of atherosclerosis and is associated with plaque rupture and occlusion of the vessel;2)calcification of media layer, or Mockenberg's sclerosis, is observed in both capacitance vessels and in muscular vessels, it causes arterial stiffness and an high pulse pressure, and is an independent risk factor for mortality of ESRD patients.

Both types of calcifications have an important impact in terms of morbidity and mortality in patients with ESRD especially if the calcification pattern affects the coronary arteries.

It is often difficult to evaluate if the calcification process is mainly located in the intima, in the media or in both. New imaging techniques have recently been used in order to reliably detect and objectively measure the extent of vascular calcification. These techniques include the use of electron beam computed tomography (EBCT) and MSCT to quantify coronary artery calcification (CAC).

The degree of calcification within the coronary arteries is measured to obtain a calcium score. Recently, several studies have analyzed the correlation between VC inhibitors and promoters and both cardiovascular disease and VC . In particular, these studies have analysed the role of fetuin A, MGP, OPG, OPN. Just few studies involved uremic patients and they considered only some of these inhibitory factors individually.

The aim of our study is to evaluate in a cohort of 253 patients, the possible associations of CAC score assessed by MSCT with risk factors of VC.

We selected 253 chronic hemodialysis patients among those undergoing hemodialysis at the Nephrology Dialysis and Renal Transplantation Unit, S.Orsola University Hospital, Bologna, Italy between April 2003 and March 2008. All the patients started dialysis from at least 6 months at the beginning of the study. All the patients are considered for gender, age on starting dialysis, months of hemodialysis, length of the period starting from the chronic renal failure onset to the beginning of dialysis, BMI, blood arterial pressure, tobacco abuse.

The mean age is 62.5 ± 13.5 years, the mean dialysis age is 41.6 ± 62.8 months. For each patient a blood sample is drawn to check the basal values of hemoglobin, hematocrit, folates, vitamin B12, C reactive protein, PTH, calcium, phosphorus, albumin, alkaline phosphatase, total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides, uric acid, fibrinogen, homocysteine. To better understand the mineral metabolism TGFb1, fetuin A, OPG, FGF 23, OPN and MGP will be checked. The values for each patient will be the median of 4 determinations, each sample was drawn before the midweek dialysis session. The period of exposure to a calcium phosphate product major than 55 mg/dl is also evaluated in all the patients (days CaxP>55). For this measure the maximum phosphate value is considered, for those patients who assume calcium based phosphate binders the measure of calcium phosphate product is obtained considering the period of maximum oral assumption of these drugs. Furthermore the calcium phosphate product is assessed monthly, in the period of dialysis before the beginning of the study, and the times when the measure exceeded 55 mg/dl (n CaxP >55) are recorded.

In the same way is assessed the period of exposure to a phosphate concentration > 6 mg/dl and the times when the marker exceeded 6 mg/dl.

The kind of phosphate binders is recorded focusing on the different associations between the drugs commercially available. The cardiovascular status of the patient is more strictly defined with a score ranging from 0 to 2 for each patient: 0 is the absence of any cardiovascular event in the patient clinical history, 1 as one VC event, 2 as two or more cardiovascular event. As regards the cardiovascular diseases screening, it is evaluated as follows: presence or absence of ischemic cardiomyopathy, cerebral or peripheral vasculopathy. Coronary artery disease was checked by means of one of the following parameters: 1) previous documentation of acute myocardial infarction; 2) symptomatic VC events in the clinical history confirmed by a positive treadmill test; 3) coronary artery stenosis more than 50% in one of the three major coronary vessels documented by an angiographic study. Cerebrovascular disease was investigated by one of the following criteria: 1) a previous ictus cerebri; b) carotid vessel stenosis more than 50% documented by a Doppler exam. Peripheral vascular disease was assessed by the evidence of claudication intermittens, previous surgical procedure, angiographic or Doppler documentation of significative stenosis in abdominal, iliac and femoral vessels.

All the patients undergo to MSCT for the determination of coronary vascular calcification and the assessment of the calcium score. Instrumental evaluation of coronary vascular calcification and the quantification of the coronary calcium score is obtained by means of Somatom Sensation 16 Cardiac (Siemens Farcheim, Germany), the calcium score was assessed by means of a specific software (Syngo Ca-score, Siemens) according to the Agatston system (18).

Patients are also grouped by means of member of cardiovascular events and by means of serum biochemistry for bone turnover to assess if any difference might emerge. A further group of patients was obtained for BMI dividing patients with BMI < 18.5, with BMI between 18.5 and 30 and over 30 to consider any possible difference of calcium score.

ELIGIBILITY:
Inclusion Criteria:

* All the patients have started dialysis from at least 6 months

Exclusion Criteria:

* Recent infectious or cardiovascular disease in the last month before the enrollment in the study;
* Malignancies;
* Active bleeding;
* Therapy with ace inhibitors or angiotensin II blocking drugs;
* Enrollment in other study protocols;
* Bone fractures in the last year;
* Paget's disease;
* Bisphosphonate therapy.
* Inflammation active process

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 253 chronic hemodialysis patients were selected among those undergoing hemodialysis at the Nephrology Dialysis and Renal Transplantation Unit, S.Orsola University Hospital, Bologna, Italy between April 2003 and March 2008. All the patients have started dialysis from at least 6 months at the beginning of the study.
Sampling Method: Probability Sample
Enrollment: 253 (Actual)
Dates: Start 2004-11; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
The aim of our study was to evaluate in a cohort of 253 patients, the possible associations of CAC score assessed by MSCT with risk factors of VC. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Stefoni, Professor, Study Director — St.Orsola Malpighi University Hospital
Locations (1):
- Nhephrology Dialysis Transplantation Unit St.Orsola University Hospital, Bologna, Italy

REFERENCES:
- [Background] Go AS, Chertow GM, Fan D, McCulloch CE, Hsu CY. Chronic kidney disease and the risks of death, cardiovascular events, and hospitalization. N Engl J Med. 2004 Sep 23;351(13):1296-305. doi: 10.1056/NEJMoa041031. PMID 15385656
- [Background] Moe SM, Chen NX. Pathophysiology of vascular calcification in chronic kidney disease. Circ Res. 2004 Sep 17;95(6):560-7. doi: 10.1161/01.RES.0000141775.67189.98. PMID 15375022
- [Background] Goodman WG, London G, Amann K, Block GA, Giachelli C, Hruska KA, Ketteler M, Levin A, Massy Z, McCarron DA, Raggi P, Shanahan CM, Yorioka N; Vascular Calcification Work Group. Vascular calcification in chronic kidney disease. Am J Kidney Dis. 2004 Mar;43(3):572-9. doi: 10.1053/j.ajkd.2003.12.005. No abstract available. PMID 14981617
- [Background] Giachelli CM. Vascular calcification mechanisms. J Am Soc Nephrol. 2004 Dec;15(12):2959-64. doi: 10.1097/01.ASN.0000145894.57533.C4. PMID 15579497
- [Background] El-Abbadi M, Giachelli CM. Mechanisms of vascular calcification. Adv Chronic Kidney Dis. 2007 Jan;14(1):54-66. doi: 10.1053/j.ackd.2006.10.007. PMID 17200044
- [Background] Jono S, Shioi A, Ikari Y, Nishizawa Y. Vascular calcification in chronic kidney disease. J Bone Miner Metab. 2006;24(2):176-81. doi: 10.1007/s00774-005-0668-6. PMID 16502129
- [Background] Collin-Osdoby P. Regulation of vascular calcification by osteoclast regulatory factors RANKL and osteoprotegerin. Circ Res. 2004 Nov 26;95(11):1046-57. doi: 10.1161/01.RES.0000149165.99974.12. PMID 15564564
- [Background] Schwarz U, Buzello M, Ritz E, Stein G, Raabe G, Wiest G, Mall G, Amann K. Morphology of coronary atherosclerotic lesions in patients with end-stage renal failure. Nephrol Dial Transplant. 2000 Feb;15(2):218-23. doi: 10.1093/ndt/15.2.218. PMID 10648668
- [Background] London GM. Cardiovascular calcifications in uremic patients: clinical impact on cardiovascular function. J Am Soc Nephrol. 2003 Sep;14(9 Suppl 4):S305-9. doi: 10.1097/01.asn.0000081664.65772.eb. PMID 12939386
- [Background] Goodman WG, Goldin J, Kuizon BD, Yoon C, Gales B, Sider D, Wang Y, Chung J, Emerick A, Greaser L, Elashoff RM, Salusky IB. Coronary-artery calcification in young adults with end-stage renal disease who are undergoing dialysis. N Engl J Med. 2000 May 18;342(20):1478-83. doi: 10.1056/NEJM200005183422003. PMID 10816185
- [Background] Raggi P, Boulay A, Chasan-Taber S, Amin N, Dillon M, Burke SK, Chertow GM. Cardiac calcification in adult hemodialysis patients. A link between end-stage renal disease and cardiovascular disease? J Am Coll Cardiol. 2002 Feb 20;39(4):695-701. doi: 10.1016/s0735-1097(01)01781-8. PMID 11849871
- [Background] Braun J, Oldendorf M, Moshage W, Heidler R, Zeitler E, Luft FC. Electron beam computed tomography in the evaluation of cardiac calcification in chronic dialysis patients. Am J Kidney Dis. 1996 Mar;27(3):394-401. doi: 10.1016/s0272-6386(96)90363-7. PMID 8604709
- [Background] Blacher J, Guerin AP, Pannier B, Marchais SJ, London GM. Arterial calcifications, arterial stiffness, and cardiovascular risk in end-stage renal disease. Hypertension. 2001 Oct;38(4):938-42. doi: 10.1161/hy1001.096358. PMID 11641313
- [Background] Agatston AS, Janowitz WR, Hildner FJ, Zusmer NR, Viamonte M Jr, Detrano R. Quantification of coronary artery calcium using ultrafast computed tomography. J Am Coll Cardiol. 1990 Mar 15;15(4):827-32. doi: 10.1016/0735-1097(90)90282-t. PMID 2407762
- [Background] Jahnen-Dechent W, Schafer C, Ketteler M, McKee MD. Mineral chaperones: a role for fetuin-A and osteopontin in the inhibition and regression of pathologic calcification. J Mol Med (Berl). 2008 Apr;86(4):379-89. doi: 10.1007/s00109-007-0294-y. Epub 2007 Dec 15. PMID 18080808
- [Background] Ix JH, Chertow GM, Shlipak MG, Brandenburg VM, Ketteler M, Whooley MA. Association of fetuin-A with mitral annular calcification and aortic stenosis among persons with coronary heart disease: data from the Heart and Soul Study. Circulation. 2007 May 15;115(19):2533-9. doi: 10.1161/CIRCULATIONAHA.106.682450. Epub 2007 May 7. PMID 17485576
- [Background] Dhore CR, Cleutjens JP, Lutgens E, Cleutjens KB, Geusens PP, Kitslaar PJ, Tordoir JH, Spronk HM, Vermeer C, Daemen MJ. Differential expression of bone matrix regulatory proteins in human atherosclerotic plaques. Arterioscler Thromb Vasc Biol. 2001 Dec;21(12):1998-2003. doi: 10.1161/hq1201.100229. PMID 11742876
- [Background] Scatena M, Liaw L, Giachelli CM. Osteopontin: a multifunctional molecule regulating chronic inflammation and vascular disease. Arterioscler Thromb Vasc Biol. 2007 Nov;27(11):2302-9. doi: 10.1161/ATVBAHA.107.144824. Epub 2007 Aug 23. PMID 17717292
- [Background] Ketteler M, Bongartz P, Westenfeld R, Wildberger JE, Mahnken AH, Bohm R, Metzger T, Wanner C, Jahnen-Dechent W, Floege J. Association of low fetuin-A (AHSG) concentrations in serum with cardiovascular mortality in patients on dialysis: a cross-sectional study. Lancet. 2003 Mar 8;361(9360):827-33. doi: 10.1016/S0140-6736(03)12710-9. PMID 12642050
- [Result] Foley RN, Parfrey PS, Sarnak MJ. Epidemiology of cardiovascular disease in chronic renal disease. J Am Soc Nephrol. 1998 Dec;9(12 Suppl):S16-23. PMID 11443763
- [Result] Sarnak MJ, Levey AS, Schoolwerth AC, Coresh J, Culleton B, Hamm LL, McCullough PA, Kasiske BL, Kelepouris E, Klag MJ, Parfrey P, Pfeffer M, Raij L, Spinosa DJ, Wilson PW; American Heart Association Councils on Kidney in Cardiovascular Disease, High Blood Pressure Research, Clinical Cardiology, and Epidemiology and Prevention. Kidney disease as a risk factor for development of cardiovascular disease: a statement from the American Heart Association Councils on Kidney in Cardiovascular Disease, High Blood Pressure Research, Clinical Cardiology, and Epidemiology and Prevention. Circulation. 2003 Oct 28;108(17):2154-69. doi: 10.1161/01.CIR.0000095676.90936.80. No abstract available. PMID 14581387
- [Result] Kalantar-Zadeh K, Ikizler TA, Block G, Avram MM, Kopple JD. Malnutrition-inflammation complex syndrome in dialysis patients: causes and consequences. Am J Kidney Dis. 2003 Nov;42(5):864-81. doi: 10.1016/j.ajkd.2003.07.016. PMID 14582032